CLINICAL TRIAL: NCT05443906
Title: Study of Adapted Exercise and Mindfulness Interventions to Improve Motor Function and Sleep Quality in Individuals with Neurodegenerative Disease
Brief Title: Home Exercise for Individuals with Neurodegenerative Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Principal Investigator, jennifer keller, Physical Therapist, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JHSOM_IRB00309985
Record Dates: First submitted 2022-05-11; First posted 2022-07-05 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Neurodegenerative Diseases; Leukodystrophy; Ataxia; LBSL; Leukoencephalopathy with Brain Stem and Spinal Cord Involvement and High Lactate Syndrome (Disorder); Leukoencephalopathy with Brainstem and Spinal Cord Involvement and Lactate Elevation; Cerebellar Ataxia; Adrenomyeloneuropathy
MeSH Terms: conditions — Neurodegenerative Diseases; Ataxia; Leukoencephalopathy with Brainstem and Spinal Cord Involvement and Lactate Elevation; Cerebellar Ataxia; Adrenoleukodystrophy

STUDY DESIGN:
Intervention Model Description: Pre-test post-test design. Based on pre-test assessments participants will be instructed in an individualized exercise program. Participants will participate in 18 hours of remotely supervised and home practice exercises.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Home exercise (Experimental): Individually designed home exercise program
  Interventions: Behavioral: Home exercise

INTERVENTIONS:
Behavioral: Home exercise — Exercise to address limitations impacting walking

SUMMARY:
The primary goal of this study is to address the need for targeted therapeutic interventions for impairments that impact walking in related neurodegenerative diseases.

DETAILED DESCRIPTION:
This study will inform clinicians in quantitatively assessing baseline disease severity, selectively applying the appropriate exercise to the disease pathology, and measuring efficacy of the exercise intervention.

As part of this overall goal, the aims are to:

A. Determine feasibility of remotely supervised exercise programs. B. Optimize remote outcome measures for clinical monitoring and towards future clinical trials.

C. Measure changes in balance and walking post intervention.

ELIGIBILITY:
Inclusion Criteria:

* The eligibility criteria for males is X-linked adrenoleukodystrophy as determined by biochemical determination or genetic testing.
* The eligibility criteria for females is X-linked adrenoleukodystrophy as determined by biochemical determination, genetic testing, or pedigree analysis.
* The Leukoenceophalopathy with brainstem and spinal cord involvement and lactate elevation inclusion criterion is a confirmed DARS2 mutation through genetic analysis.
* For people with cerebellar ataxia, people with diagnoses of cerebellar damage from stroke, tumor or degeneration will be included. Those with a genetically confirmed cerebellar disorder will be asked to provide their genetic testing to note their particular type of ataxia.
* We will also include patients with other neurodegenerative diseases similar to these disorders as determined by chart review and clinical exam.

Healthy Volunteers

* Able to stand for 30 seconds without upper extremity support
* Ambulatory (including use of a cane or a walker)
* Able to walk for 2 minutes

Exclusion Criteria:

* Other medical or psychological conditions which in the clinical judgement of the investigator would interfere with acquiring the study information or performing the exercises safely including but not limited to:

Uncontrolled hypertension, orthopedic conditions, diabetes, seizure disorder, peripheral vestibular loss, severe aphasia, dementia, pregnancy

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in NeuroQOL lower extremity | baseline 12 weeks
  Patient reported outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Keller, PT, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No